CLINICAL TRIAL: NCT05933733
Title: A Prospective Registry Study to Evaluate Oncologic Outcomes and Toxicities of Salvage Treatment in Patients With Locoregionally Recurrent Breast Cancer
Brief Title: Oncologic Outcomes and Toxicities of Salvage Treatment in Patients With Locoregionally Recurrent Breast Cancer
Acronym: SALT-LRR
Status: Recruiting | Type: Observational
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Haeyoung Kim, Associate Professor, Samsung Medical Center
Other Study IDs: 2023-05-023
Record Dates: First submitted 2023-06-27; First posted 2023-07-06 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Salvage Therapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Residual tissue archived at the pathology department after histologic confirmation of diagnosis
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Salvage treatment after locoregional recurrence: Participants who previously completed standard treatment for breast cancer and experienced locoregional recurrence alone will be undergo salvage treatment including surgery and/or radiation therapy.
  Interventions: Other: Salvage treatment (surgery and/or radiation therapy)

INTERVENTIONS:
Other: Salvage treatment (surgery and/or radiation therapy) — Appropriate salvage treatment (surgery and/or radiation therapy) will be selected by the treating clinicians considering the disease status.

SUMMARY:
The purpose of this study is to evaluate clinical outcomes and adverse events of salvage treatment for locoregional recurrence of breast cancer.

The main questions it aims to answer are:

* Clinical outcomes after salvage treatment for locoregional recurrence
* Adverse events and quality of life after salvage treatment for locoregional recurrence
* Patient characteristics and treatment specifics which are related to the clinical outcomes and/or adverse events
* Molecular signature associated with treatment resistance

Participants will be assessed by multi-dimensional methods during and after radiation therapy:

* Assessment for the disease status (disease-free or recurrence) including physical and radiologic examination
* Assessment for the adverse events according to CTCAE version 5.0
* Assessment for the molecular signature using residual tissue after pathologic diagnosis
* Assessment for the quality of life using questionnaires (BREAST-Q)

ELIGIBILITY:
Inclusion Criteria:

* Female patients with age 18 to 100.
* Previous standard definitive treatment for initial breast cancer
* Locoregional recurrence without distant metastasis
* Planned salvage treatment for locoregional recurrence
* Informed consent of the participant

Exclusion Criteria:

- Not anticipated for complying the study protocol

Ages: 18 Years to 100 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Breast cancer patients who underwent standard treatment for initial breast cancer and experienced locoregional recurrence without distant metastasis which is eligible for salvage treatment can be enrolled for this study.
Sampling Method: Non-Probability Sample
Enrollment: 190 (Estimated)
Dates: Start 2023-07-04 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2033-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival | 5 years from the initiation of the salvage therapy
  The event for progression-free survival was defined as any disease progression or breast cancer-related death.
Rate of adverse events | 5 years from the initiation of the salvage therapy
  Adverse events related to the salvage therapy will be reported and incidence rate will be calculated.

SECONDARY OUTCOMES:
Locoregional failure rate | 5 years from the initiation of the salvage therapy
  The event for locoregional failure rate was defined as recurrence in breast / chest wall or regional lymph node area.
Cancer-specific survival | 5 years from the initiation of the salvage therapy
  The event for cancer-specific survival was defined as death of the participant related to the breast cancer.
Quality of life (BREAST-Q) | 5 years from the initiation of the salvage therapy
  Quality of life of the participants will be evaluated according to the BREAST-Q™ questionnaires. Higher Q-Score indicates better quality of life.
Breast cosmesis | 5 years from the initiation of the salvage therapy
  Cosmesis of the breast will be evaluated according to Harvard/National Surgical Adjuvant Breast and Bowel Project (NSABP)/Radiation Therapy Oncology Group (RTOG) Breast Cosmesis grading scale. This is a 4-point scale (Excellent, Good, Fair, and Poor), and evaluated by the clinicians.

CONTACTS AND LOCATIONS:
Overall Officials: Haeyoung Kim, Principal Investigator — Samsung Medical Center
Locations (1):
- Samsung Medical Center, Seoul, South Korea